CLINICAL TRIAL: NCT07067359
Title: Effect of Intensive Nutrition Intervention in Esophagogastric Cancer Patients With Neoadjuvant Therapy: A Randomized Clinical Trial
Brief Title: The Intensive Nutritional Support in Esophageal Cancer Undergoing Neoadjuvant Therapy
Acronym: INSECNT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Clinical Professor, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX2023382
Record Dates: First submitted 2025-01-23; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; nutrition; Neoadjuvant therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Enteral Nutrition; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Experimental: Intensive Nutrition therapy (INT) Esophageal cancer patients with nutritional risk undergoing neoadjuvant therapy received dietary guidance and necessary nutritional supplements during hospitalization. In addition to this, they continued to receive ongoing nutritional counseling and monitoring after discharge to ensure sustained nutritional support.
  Active Comparator: Standard Nutrition Therapy (SNT) Esophageal cancer patients with nutritional risk undergoing neoadjuvant therapy received a conventional nutritional support regimen during hospitalization, including dietary guidance and necessary nutritional supplements.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Nutrition therapy (INT) (Experimental): Esophageal cancer patients with nutritional risk undergoing neoadjuvant therapy received dietary guidance and necessary nutritional supplements during hospitalization. In addition to this, they continued to receive ongoing nutritional counseling and monitoring after discharge to ensure sustained nutritional support.
  Interventions: Dietary Supplement: Enteral Nutrition
- Standard Nutrition Therapy (SNT) (Active Comparator): Esophageal cancer patients with nutritional risk undergoing neoadjuvant therapy received a conventional nutritional support regimen during hospitalization, including dietary guidance and necessary nutritional supplements.
  Interventions: Dietary Supplement: Enteral Nutrition

INTERVENTIONS:
Dietary Supplement: Enteral Nutrition — This study selected patients with esophageal cancer undergoing neoadjuvant therapy as the research subjects. All enrolled patients underwent comprehensive nutritional risk screening and malnutrition assessment prior to enrollment. After the completion of nutritional risk screening and assessment, patients identified with nutritional risk were randomly assigned to two groups: the Standard Nutrition Therapy group (SNT) and the Intensive Nutrition Therapy group (INT). Patients in the SNT group received a conventional nutritional support regimen during hospitalization, which included dietary guidance and necessary nutritional supplements. In addition to the standard regimen, patients in the INT group continued to receive ongoing nutritional counseling and nutritional supplement support after discharge to ensure sustained nutritional support.
  Other Names: Nutritional supplements; Dietary guidance

SUMMARY:
Patients with esophageal cancer undergoing neoadjuvant therapy were selected as research subjects for nutritional risk screening and malnutrition assessment. Patients identified with nutritional risk were randomized into the standard nutrition therapy group (SNT) and the intensive nutrition therapy group (INT). The surgical rate was evaluated in both groups of patients, and the effects of nutritional support therapy on nutritional status and quality of life were investigated.

DETAILED DESCRIPTION:
Esophageal cancer is one of the most common malignant tumors in China, with high incidence and mortality rates. Due to its anatomical location and pathological characteristics, patients with esophageal cancer often experience symptoms such as dysphagia and reduced appetite at an early stage of the disease, leading to inadequate nutritional intake and subsequent malnutrition. Malnutrition not only weakens the immune function of patients but also reduces their tolerance to surgery, radiotherapy, and chemotherapy. It may also prolong hospital stays, increase the incidence of complications, and ultimately affect patient prognosis and quality of life. Therefore, conducting nutritional risk screening and malnutrition assessment for patients with esophageal cancer, and providing targeted nutritional support therapy based on these assessments, is of significant importance for improving clinical outcomes.

This study selected patients with esophageal cancer undergoing neoadjuvant therapy as the research subjects. All enrolled patients underwent comprehensive nutritional risk screening and malnutrition assessment prior to enrollment. After completing the nutritional risk screening and assessment, patients identified with nutritional risk were randomly divided into two groups: the Standard Nutrition Therapy group (SNT) and the Intensive Nutrition Therapy group (INT). Patients in the Standard Nutrition Therapy group (SNT) received a conventional nutritional support regimen during hospitalization, which included dietary guidance and necessary nutritional supplements. In contrast, patients in the Intensive Nutrition Therapy group (INT) not only received the standard regimen but also continued to receive ongoing nutritional counseling and monitoring after discharge, ensuring sustained nutritional support for the patients.

The primary research content of this study includes the surgical resection rate. By comparing the surgical rates between the two groups of patients, the impact of different nutritional support regimens on patients' surgical opportunities was assessed. Additionally, the effectiveness of nutritional support therapy in improving patients' nutritional status was evaluated by regularly monitoring changes in nutritional indicators such as body weight, body mass index (BMI), and serum albumin levels.

This study aims to provide high-quality clinical evidence for the nutritional support treatment of patients with esophageal cancer through a randomized controlled trial. We anticipate that patients in the intensive nutrition therapy group will outperform those in the standard nutrition therapy group in terms of surgical rates and improvement in nutritional status. Through this study, we hope to further optimize the nutritional management strategies for patients with esophageal cancer, provide more targeted nutritional support regimens for clinicians, and thereby improve patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Esophageal cancer；
2. Patients were staged as cT1b-cT2N+M0 or cT3-cT4a, any N, M0. Based on the location of the tumor and clinical staging, they were defined as locally advanced resectable esophageal cancer；
3. Patients planned for neoadjuvant therapy, with radical surgical resection intended after neoadjuvant treatment；
4. Normal gastrointestinal function；
5. PG-SGA score >3;
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2分.

Exclusion Criteria:

1. Other tumors, including pancreatic cancer, liver cancer and other solid digestive tract tumors, colon cancer, rectal cancer and other tubular lower digestive tract tumors;
2. Have serious heart, lung and brain diseases;
3. Patients with unstable vital signs and multiple organ failure;
4. The patient has poor cognitive ability and is unable to answer questions or fill out questionnaires;
5. Eastern Cooperative Oncology Group score >2;
6. The investigator believes that the subjects have a history of other serious systemic diseases or are not suitable for participating in this clinical study for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Surgical resection rate | Through study completion, an average of 1 year
  The proportion of esophageal cancer patients who undergo radical surgical resection after neoadjuvant therapy.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the start of the first neoadjuvant treatment to four weeks after the first tumor assessment.
  The Objective Response Rate (ORR) refers to the proportion of patients whose tumor lesions completely disappear (Complete Response, CR) or partially shrink (Partial Response, PR) during neoadjuvant therapy.
The rate of pathological complete response (pCR) | Through study completion, an average of 1 year
  Pathological Complete Response (pCR) refers to the absence of any residual cancer cells in the tumor tissue resected after neoadjuvant therapy.
Event free survival (EFS) | From the start of the first neoadjuvant treatment, the observation period is up to 2 years.
  Event-Free Survival (EFS) refers to the time from the start of treatment to the first occurrence of disease progression, recurrence, death, or other predefined adverse events.
Overall survival (OS) | From the start of the first neoadjuvant treatment, the observation period is up to 2 years.
  Overall Survival (OS) refers to the time from the start of treatment to the patient's death from any cause.
Nutrition status | Perioperative
  The nutritional status of patients was assessed using Patient-Generated Subjective Global Assessment (PG-SGA) before neoadjuvant therapy and before surgery. PG-SGA is a multidimensional tool for assessing patients' nutritional status and is widely used in oncology and other chronic catabolic diseases. This tool combines the patient's self-assessment with the assessment by healthcare professionals and can comprehensively reflect the patient's nutritional state and nutritional risk. The higher the score, the worse the patient's nutritional status. 0-1 point: Good nutritional status. 2-8 points: Suspected or moderate malnutrition. ≥9 points: Severe malnutrition.
Quality of life (QOL) | Perioperative
  Quality of life was assessed before neoadjuvant therapy and before surgery. Quality of life was assessed using the Uropean Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale. The EORTC QLQ-C30 scale is a standardized and validated tool for assessing health-related quality of life (HRQoL) in cancer patients, developed by the European Organization for Research and Treatment of Cancer (EORTC). Scoring range: 0-100 points. Higher scores indicate better functional status and higher quality of life.